CLINICAL TRIAL: NCT05588869
Title: Cyclosporine Adverse Outcomes in Steroid Dependent and Frequent Relapsing Nephrotic Syndrome in Children;Single Center Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Talaat Mahmoud Abdelaal, resident doctor at pediatric department, Sohag University
Other Study IDs: Soh-Med-22-10-01
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Steroid Dependent and Frequent Relapsing Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation of the adverse outcomes of Cyclosporine in steroid dependent and frequent relapsing nephrotic syndrome in children — The interventions that will be done include collection of the following data : age at disease onset, disease duration, type of steroid response, age at the start of CsA treatment, dose and duration of CsA treatment, mean values of the maintenance doses of CsA and their trough blood levels and observation of the side effects. serum creatinine at regular intervals before and after CsA treatment and renal biopsy for those who are on CsA for more than 2-3 years would be done.

SUMMARY:
Nephrotic syndrome (NS) is the most common glomerular disorder in children with significant morbidity and mortality and affects about 1-3 per 100,000 children aged below 16 years. Nephrotic syndrome is characterized by the presence of edema, proteinuria: uPCR (urine protein creatinine ratio) ≥200 mg/mmol (≥2 g/g) or 3+ protein on urine dipstick and hypoalbuminemia less than 3 g/dl).Nephrotic syndrome is classified according to response to steroids into steroid sensitive and steroid resistant. Approximately 90% of all cases are steroid-sensitive with an initial episode successfully treated with a standardized treatment protocol of steroids. However, about 80% of these patients experience further relapses. Of these, 50% are steroid dependent and frequent relapsers. While any relapse can be treated with steroids, children may be vulnerable to the side effects of a high cumulative dose of steroids such as obesity, growth impairment, behavioral alterations and attention problems, as well as reduced quality of life and family stress. To minimize steroid toxicity in patients with steroid-dependent and frequently relapsing nephrotic syndrome, a number of immunosuppressive agents are recommended as maintenance therapeutic agents. Among those are cyclosporine A, tacrolimus, mycophenolate mofetil (MMF), cyclophosphamide, levamisole and rituximab. Cyclosporin-A (CsA) is a calcineurin inhibitor that is well recognized as having a steroid sparing effect in steroid-dependent and frequently relapsing NS and has a role in the maintenance of complete remission in more than 75% of patients with SDNS during discontinuation of steroids. However, early withdrawl of cysclosporine may lead to relapses so the patient may be dependent on cyclosporine for years. The long-term use of CsA has been identified to be a risk factor of unsatisfactory effects such as nephrotoxicity, hypertension and cosmetic symptoms such as (gum hypertrophy and hirsutism). Therefore, close observation of the side effects of cyclosporine is very important as well as regular follow up of blood pressure and kidney function tests. Also, estimation of trough blood levels of CsA is required in patients with suspected non compliance, unsatisfactory response or nephrotoxicity (increase in serum creatinine by 30% or more from the baseline) aiming for the lowest levels that maintain remission and avoid toxicity (target 12-hr trough level of 60-150 ng/ml). Kidney biopsy could be included as a component of the long-term CsA protocol to test for CsA-associated nephropathy if given more than 2-3 years. CsA nephrotoxicity is primarily caused by chronic ischemic insult to the kidney, resulting in arteriolar hyalination and tubulointerstitial changes, including striped interstitial fibrosis, tubular vacuolization, and atrophy.The aim of this study is to determine the adverse outcomes of Cyclosporine in children with steroid dependent and frequent relapsing nephrotic syndrome in Sohag University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* The study will include children and adolescents diagnosed as steroid dependent and frequent relapsing nephrotic syndrome with disease onset from one to fifteen years and treated with cyclosporine A in the Paediatric nephrology clinic, Sohag University Hospital

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children and adolescents diagnosed as steroid dependent and frequent relapsing nephrotic syndrome with disease onset from one to fifteen years and treated with cyclosporine A in the Paediatric nephrology clinic, Sohag University Hospital
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-10-20 (Estimated); Primary Completion 2023-04-20 (Estimated); Study Completion 2023-04-20 (Estimated)

PRIMARY OUTCOMES:
observation of the side effects of cyclosporine in steroid dependent and frequent relapsing nephrotic syndrome in children | 6 months
  observation and follow up of unsatisfactory effects of cyclosporine such as nephrotoxicity, hypertension and cosmetic symptoms such as (gum hypertrophy and hirsutism).serum creatinine at regular intervals before and after CsA treatment, renal biopsy for those who are on CsA for more than 2-3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Glomerular Diseases Work Group. KDIGO 2021 Clinical Practice Guideline for the Management of Glomerular Diseases. Kidney Int. 2021 Oct;100(4S):S1-S276. doi: 10.1016/j.kint.2021.05.021. No abstract available. PMID 34556256
- [Background] Ehren R, Benz MR, Brinkkotter PT, Dotsch J, Eberl WR, Gellermann J, Hoyer PF, Jordans I, Kamrath C, Kemper MJ, Latta K, Muller D, Oh J, Tonshoff B, Weber S, Weber LT; German Society for Pediatric Nephrology. Pediatric idiopathic steroid-sensitive nephrotic syndrome: diagnosis and therapy -short version of the updated German best practice guideline (S2e) - AWMF register no. 166-001, 6/2020. Pediatr Nephrol. 2021 Oct;36(10):2971-2985. doi: 10.1007/s00467-021-05135-3. Epub 2021 Jun 6. PMID 34091756
- [Background] Kuroyanagi Y, Gotoh Y, Kasahara K, Nagano C, Fujita N, Yamakawa S, Yamamoto M, Takeda A, Uemura O. Effectiveness and nephrotoxicity of a 2-year medium dose of cyclosporine in pediatric patients with steroid-dependent nephrotic syndrome: determination of the need for follow-up kidney biopsy. Clin Exp Nephrol. 2018 Apr;22(2):413-419. doi: 10.1007/s10157-017-1444-3. Epub 2017 Jul 11. PMID 28699031
- [Background] Hampson KJ, Gay ML, Band ME. Pediatric Nephrotic Syndrome: Pharmacologic and Nutrition Management. Nutr Clin Pract. 2021 Apr;36(2):331-343. doi: 10.1002/ncp.10622. Epub 2021 Jan 19. PMID 33469930